CLINICAL TRIAL: NCT01215474
Title: Pathomolecular Analysis of Rare EGFR Mutations in Advanced NSCLC
Status: Completed | Type: Observational
Sponsor: Provitro GmbH (Industry)
Collaborators: AstraZeneca (Industry); Charite University, Berlin, Germany (Other)
Other Study IDs: AZ-NSCLC 18+
Record Dates: First submitted 2010-10-05; First posted 2010-10-06 (Estimated); Last update posted 2011-06-16 (Estimated); Status verified 2010-10

CONDITIONS: Mutations in Exons 18 to 21

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- NSCLC Stadium III-IV

SUMMARY:
While current mutational analyses comprise exons 19 and 21 in which the majority of EGFR-mutations occur, this study aims at investigating the relevance of exon 18 and 20 mutations. Therefore, the investigators analyse 500 routine tumor samples with respect to the above mentioned exons and correlate the results to the clinical outcome. This approach will enable us to potentially identify patients that might in the future benefit from targeted therapy (EGFR-inhibition).

ELIGIBILITY:
Inclusion Criteria:

* NSCLC Stadium III-IV

Exclusion Criteria:

* no NSCLC or different stadium

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who were biopsied and/or received surgery for NSCLC diagnostics
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Pathology, Charité University Medicine Berlin, Berlin, Germany